CLINICAL TRIAL: NCT02387385
Title: Hypothermia for Encephalopathy in Low and Middle-Income Countries Trial
Acronym: HELIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thayyil, Sudhin (Individual)
Collaborators: Madras Medical College (Other Government); Indira Gandhi Medical College, Shimla (Other); Lokmanya Tilak Municipal Medical College and Hospital (Other); Imperial College London (Other); Maulana Azad Medical College (Other); Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other); University of Kelaniya (Other); Medical College Trivandrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15HH
Record Dates: First submitted 2015-02-27; First posted 2015-03-13 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Neonatal Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Whole body cooling to 33 degrees C to 34 degrees C
  Interventions: Device: Whole body cooling (Tecotherm)
- Standard of Care (No Intervention): Standard of care

INTERVENTIONS:
Device: Whole body cooling (Tecotherm) — Whole body cooling to 33 to 34 C using Tecotherm
  Arms: Intervention

SUMMARY:
Neonatal Encephalopathy is a serious condition arising from unexpected lack of cerebral blood flow and oxygen supply to the foetal brain at the time of birth. Every year, approximately one million babies die from neonatal encephalopathy in low and middle-income countries and a quarter of these deaths occur in India.

In the past decade, a number of clinical trials in high-income countries has shown that cooling therapy along with optimal neonatal intensive care reduces death and neurodisability after neonatal encephalopathy. Cooling therapy is now used as a standard therapy after neonatal encephalopathy in all high income countries, including the UK.

Although the burden of neonatal encephalopathy is far higher in low and middle-income countries, the safety and efficacy data on cooling therapy from high income cooling trials cannot be extrapolated to these settings, due to the difference in population co-morbidities and sub-optimal neonatal intensive care.

The HELIX trial proposes to examine whether whole body cooling to 33.5°C initiated within 6 hours of birth and continued for 72 hours reduces death or neurodisability at 18 months after neonatal encephalopathy in public sector neonatal units in India.

A total of 408 babies with moderate or severe neonatal encephalopathy will be recruited from the participating centres in India over an 18 to 24 month period. The babies will be randomly allocated to whole body cooling or usual care. The cooling therapy will be achieved using an approved cooling device (Tecotherm) that is already in clinical use in the UK and in India. MR imaging and spectroscopy will be performed at 1 week of age to examine the brain injury. Neurodevelopmental outcomes will be assessed at 18 months of age. Primary outcome measure is death or moderate/severe neurodisability at 18 months.

DETAILED DESCRIPTION:
Although the burden of neonatal encephalopathy is far higher in low and middle-income countries, the safety and efficacy data on cooling therapy from high income cooling trials cannot be extrapolated to these settings.

Firstly, all high-income country clinical trials to date have provided cooling therapy along side optimal tertiary neonatal intensive care and cardiorespiratory support. Such tertiary care includes 1:1 expert nursing care, continuous clinical monitoring of vital physiological parameters, close attention to acid base and electrolyte balance, optimal ventilatory and inotropic support, parenteral nutrition, nitric oxide and cerebral function monitoring. These centres also have access to extra-corporeal membrane oxygenation (ECMO) facilities for infants with persistent pulmonary hypertension and meconium aspiration that may be adversely affected by cooling. The safety and efficacy of cooling therapy without optimal tertiary neonatal intensive care is unknown. Even the best resourced public sector tertiary neonatal units in India and other low and middle-income countries do not have the facilities and expertise that are comparable to the neonatal units where the high-income cooling trials were originally performed. The dangers of extrapolating the safety and efficacy data from high income country intensive care units to low and middle-income countries is well known, and has been recently re-emphasised by the increased mortality seen after fluid boluses in children with septic shock in Africa (FEAST trial). The HELIX trial will examine the safety of cooling therapy in under resourced public sector neonatal units in India, who do not have the above-mentioned facilities for providing optimal tertiary intensive care, alongside cooling therapy. Secondly, there are significant population differences in babies who suffer from encephalopathy in high-income countries and those in low and middle-income countries with a higher incidence of perinatal infection and meconium aspiration. Antenatal care is often poor, and intra uterine growth restriction and delayed hospital admission in obstructed labour are extremely common.

Thus the brain injury may be more chronic and already established, such that the window period for cooling may be already lost by the time baby is born. Two recent NICHD hypothermia workshops (2011 and 2013)14 involving experts in therapeutic hypothermia have recommended that rigorous evaluation of cooling therapy should be urgently conducted in LMIC, to ensure that the benefits of one of the most important discoveries in neonatal medicine are not lost to the population that needs it most. Without such rigorous evaluation there may be a creeping introduction of cooling therapy, which is constantly sabotaged by residual safety concerns, and it will never be widely used in India and other LMIC.

Cooling studies from low and middle-income countries A number of small randomised controlled trials have been reported from low and middle-income countries. Individual studies were small and of poor quality. The largest of these trials reported from China had excluded babies at risk of perinatal sepsis and had substantial methodological concerns. Two studies reported increased mortality with cooling. Meta-analysis of all these trials showed a trend towards reduced mortality, however this was not statistically significant (RR 0.74; 95% CI 0.4 to 1.3). More importantly, the confidence intervals were wide and therefore significant benefits or harm cannot be excluded. There were no data on long term neurological follow up after cooling therapy. In preparation for the HELIX trial, the investigators conducted a feasibility study of cooling therapy using a servo controlled cooling device (Tecotherm) in 2013/14, at Madras Medical College (MMC), Chennai. The data from 58 cooled babies with neonatal encephalopathy and 112 contemporary 'un matched' encephalopathic babies who had usual care (normothermia) admitted to the neonatal unit over a 15 month period are given below . Although the neonatal mortality in the cooled babies appears to be higher than the high-income country cooling trials, it was lower than the contemporary encephalopathic population at this hospital. High incidence of gastric bleeds and persistent metabolic acidosis were seen in both groups. The cases and controls were not matched and it is possible that the control babies were more unwell, and therefore had higher mortality (29% versus 54%; Table 1); nevertheless, these data are reassuring and support further evaluation of cooling therapy in a rigorous randomised controlled trial (manuscript in preparation). A paradox of private and public sector health care exists in India and other low and middleincome countries. Private hospitals are often very well equipped and have good tertiary intensive care facilities, but are not affordable to the low income populations. Moreover, these hospitals are relatively smaller (annual delivery rates of less than 2000), and have a low encephalopathy burden. Public sector hospitals on the other hand, tend to be much larger (20,000 to 30,000 deliveries per year) and offer free health care to the low income population. These hospitals have a huge encephalopathy burden (both inborn and out-born babies), but lack resources and good neonatal intensive care facilities. Thus, significant health benefits will occur only if the neuroprotective therapies are usable and indeed effective in public sector hospitals in the low and middle-income countries, rather than in private health care.

The HELIX trial is carefully designed to be generalizable to all under-resourced neonatal units with sub optimal neonatal intensive in India and other low and middle-income countries, that bear a very high neonatal encephalopathy burden. However, the neonatal units need to have a good quality basic neonatal care, including facilities of neonatal resuscitation, administration of intravenous fluids, drugs and basic respiratory support, but not optimal cardio respiratory or 1:1 nursing care facilities. The HELIX trial will be conducted in the real life situation of under resourced public sector neonatal units lacking optimal tertiary intensive care in India. Exclusively clinical criteria will be used for case identification and recruitment, and no laboratory parameters, neuroimaging or cerebral function monitoring will be required for eligibility. The entire cooling therapy will be provided by the existing clinical teams, and the research team will only be involved in accurate and high quality data collection, so that the trial results are reflective of the routine clinical scenario. Clearly, the population co-morbidities and resources in Indian neonatal units are different to African and other low-income country neonatal units. If the HELIX trial results suggest that cooling is safe and effective in Indian neonatal units, the next stage would be to evaluate cooling therapy in under resourced neonatal units in Africa, and other low-income countries.

The Helix trial is a two arm un-blinded pragmatic randomised controlled trial of whole body cooling versus standard care, after neonatal encephalopathy in low and middle-income countries. The investigators plan to randomise 408 babies in this trial, for which the investigators anticipate approximately 1200 babies will have to be screened for eligibility. The treatment duration (cooling therapy) is 72 hours, however the temperature of all recruited babies will be monitored during the first week after birth. Any temperature rise over >37.5°C will be active treated, both in the cooling and usual care arms, as fever increases the brain injury and adverse outcomes after neonatal encephalopathy. The neurological outcomes will be assessed between 18 to 22 months of age. The trial duration will be 4 years, consisting of a 4 week start up period, 24 month recruitment period, a 18 month follow-up period, and 5 months for data analysis and write up.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 6 hours, Birth-weight >1.8 kg, Gestation >36 weeks
2. Need for continued resuscitation at 5 minutes after birth and/or 5 minute Apgar score <6 (in babies born at hospital) or lack of cry by 5 minutes of age (for babies born at home)
3. Evidence of moderate or severe encephalopathy on clinical examination within 6 hours of age.

Exclusion Criteria:

1. Absent heart rate at 10 minute of age despite adequate resuscitation.
2. Major life threatening congenital malformation.
3. Migrant family or parents unable/unlikely to come back for follow up at 18 months.
4. Lack of parental consent.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2015-08; Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Composite outcome of Death or moderate or severe neurodisability | 18 to 22 months

SECONDARY OUTCOMES:
Mortality from any cause | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Major intracranial haemorrhage | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Gastric bleeds (fresh blood > 5 ml from nasogastric tube) | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Persistent hypotension (mean blood pressure < 40 mm of Hg requiring inotropic support) | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Pulmonary haemorrhage (Copious bloody secretions with clinical deterioration requiring change(s) in ventilatory management) | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Persistent pulmonary hypertension (Severe hypoxemia disproportionate to the severity of lung disease with a significant pre-and post ductal saturation difference on pulse oximetry) | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Prolonged blood coagulation time requiring blood products | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Culture proven early onset sepsis (isolation of a pathogenic organism from blood or cerebrospinal fluid along with clinical evidence of sepsis and elevation of C-reactive protein) | Prolonged blood coagulation time requiring blood products Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Necrotising enterocolitis (defined as abdominal distension, increased gastric aspirates and/or blood in stools together with abdominal X-ray showing bowel oedema, pneumatosis or pneumoperitoneum, i.e. Bell's staging 2 or 3) | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Cardiac arrhythmia | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Severe thrombocytopenia | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Renal failure | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Pneumonia | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Subcutaneous fat necrosis | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Duration of hospitalisation | before discharge from hospital Expected average of 3 weeks
  Expected average of 3 weeks hospital stay
Mortality | Long term (18 to 22 months)
  Expected average of 3 weeks hospital stay
Severe neurodevelopmental disability | Long term (18 to 22 months)
Microcephaly (head circumference more than 2 standard deviations below the mean) | Long term (18 to 22 months)

CONTACTS AND LOCATIONS:
Overall Officials: Sudhin Thayyil, PhD, Study Director — Imperial College London; Vania Oliveira, MSc, Principal Investigator — Imperial College London; Seetha Shankaran, MD, Principal Investigator — Wayne State University
Locations (9):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
- India (7):
  - Institute of Obstetrics and Gynaecology, Chennai, Tamil Nadu
  - Indira Gandhi Institute of Child Health, Bangalore
  - Calicut Medical College, Calicut
  - Institute of Child Health, Madras Medical College, Chennai
  - Sion Hospital, Mumbai
  - Maulana Azad Medical College, New Delhi
  - Medical College Trivandrum, Trivandrum
- University of Kelaniya, Kelaniya, Sri Lanka

REFERENCES:
- [Background] Montaldo P, Pauliah SS, Lally PJ, Olson L, Thayyil S. Cooling in a low-resource environment: lost in translation. Semin Fetal Neonatal Med. 2015 Apr;20(2):72-9. doi: 10.1016/j.siny.2014.10.004. Epub 2014 Oct 31. PMID 25457083
- [Result] Thayyil S, Oliveira V, Lally PJ, Swamy R, Bassett P, Chandrasekaran M, Mondkar J, Mangalabharathi S, Benkappa N, Seeralar A, Shahidullah M, Montaldo P, Herberg J, Manerkar S, Kumaraswami K, Kamalaratnam C, Prakash V, Chandramohan R, Bandya P, Mannan MA, Rodrigo R, Nair M, Ramji S, Shankaran S; HELIX Trial group. Hypothermia for encephalopathy in low and middle-income countries (HELIX): study protocol for a randomised controlled trial. Trials. 2017 Sep 18;18(1):432. doi: 10.1186/s13063-017-2165-3. PMID 28923118
- [Result] Thayyil S, Pant S, Montaldo P, Shukla D, Oliveira V, Ivain P, Bassett P, Swamy R, Mendoza J, Moreno-Morales M, Lally PJ, Benakappa N, Bandiya P, Shivarudhrappa I, Somanna J, Kantharajanna UB, Rajvanshi A, Krishnappa S, Joby PK, Jayaraman K, Chandramohan R, Kamalarathnam CN, Sebastian M, Tamilselvam IA, Rajendran UD, Soundrarajan R, Kumar V, Sudarsanan H, Vadakepat P, Gopalan K, Sundaram M, Seeralar A, Vinayagam P, Sajjid M, Baburaj M, Murugan KD, Sathyanathan BP, Kumaran ES, Mondkar J, Manerkar S, Joshi AR, Dewang K, Bhisikar SM, Kalamdani P, Bichkar V, Patra S, Jiwnani K, Shahidullah M, Moni SC, Jahan I, Mannan MA, Dey SK, Nahar MN, Islam MN, Shabuj KH, Rodrigo R, Sumanasena S, Abayabandara-Herath T, Chathurangika GK, Wanigasinghe J, Sujatha R, Saraswathy S, Rahul A, Radha SJ, Sarojam MK, Krishnan V, Nair MK, Devadas S, Chandriah S, Venkateswaran H, Burgod C, Chandrasekaran M, Atreja G, Muraleedharan P, Herberg JA, Kling Chong WK, Sebire NJ, Pressler R, Ramji S, Shankaran S; HELIX consortium. Hypothermia for moderate or severe neonatal encephalopathy in low-income and middle-income countries (HELIX): a randomised controlled trial in India, Sri Lanka, and Bangladesh. Lancet Glob Health. 2021 Sep;9(9):e1273-e1285. doi: 10.1016/S2214-109X(21)00264-3. Epub 2021 Aug 3. PMID 34358491
- [Result] Pant S, Elias MA, Woolfall K, Morales MM, Lincy B, Jahan I, Sumanasena SP, Ramji S, Shankaran S, Thayyil S; HELIX Trial consortium investigators. Parental and professional perceptions of informed consent and participation in a time-critical neonatal trial: a mixed-methods study in India, Sri Lanka and Bangladesh. BMJ Glob Health. 2021 May;6(5):e005757. doi: 10.1136/bmjgh-2021-005757. PMID 34020995
- [Derived] Thayyil S, Montaldo P, Krishnan V, Ivain P, Pant S, Lally PJ, Bandiya P, Benkappa N, Kamalaratnam CN, Chandramohan R, Manerkar S, Mondkar J, Jahan I, Moni SC, Shahidullah M, Rodrigo R, Sumanasena S, Sujatha R, Burgod C, Garegrat R, Mazlan M, Chettri I, Babu Peter S, Joshi AR, Swamy R, Chong K, Pressler RR, Bassett P, Shankaran S. Whole-Body Hypothermia, Cerebral Magnetic Resonance Biomarkers, and Outcomes in Neonates With Moderate or Severe Hypoxic-Ischemic Encephalopathy Born at Tertiary Care Centers vs Other Facilities: A Nested Study Within a Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2312152. doi: 10.1001/jamanetworkopen.2023.12152. PMID 37155168